CLINICAL TRIAL: NCT00552552
Title: Development and Evaluation of a Cancer-Related Fatigue Patient Education Program
Acronym: FIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bremen (Other)
Collaborators: Institute of Public Health and Nursing Research (IPP) (Unknown); German Federal Ministry of Education and Research (Other Government); Bremer Krebsgesellschaft e.V. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 41100133
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Cancer-Related Fatigue
Keywords: cancer-related fatigue; self-management; patient education; cancer survivors; chronic disease
MeSH Terms: conditions — Chronic Disease | interventions — FIBS

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Fatigue Patient Education Program (FIBS)
- 2 (Other): waiting control group
  Interventions: Behavioral: Fatigue Patient Education Program (FIBS)

INTERVENTIONS:
Behavioral: Fatigue Patient Education Program (FIBS) — 6 weekly sessions, 90 min each
  Other Names: FIBS (Fatigue individuell bewältigen - ein Selbstmanagementprogramm)
  Arms: 1
Behavioral: Fatigue Patient Education Program (FIBS) — Participation in the program after the second follow-up
  Other Names: FIBS (Fatigue individuell bewältigen - ein Selbstmanagementprogramm)
  Arms: 2

SUMMARY:
The objective of this study is to develop a structured and evidence-based self-management program to cope with cancer-related fatigue and to assess the efficacy of the intervention in cancer survivors.

DETAILED DESCRIPTION:
Background

Cancer-related fatigue (CRF) and its impact on patients quality of life has been an increasing subject of research. However, in Germany exists a lack of evidence-based interventions consistent with the multidimensional character of fatigue. The objective of this study is to develop and evaluate a self-management program for disease-free cancer patients to cope with CRF.

Methods

Based on evidence extracted from a literature review a curriculum for the self-management program was elaborated. The curriculum is currently being reviewed and validated by an expert group of oncologists, psycho-oncologists, nurses, social workers, physical therapists, health scientists, and patients. The modules will be pretested with a small number of patients, discussed in terms of feasibility and acceptance.

To determine the efficacy of the program a randomised controlled trial will be conducted: 300 patients will be allocated to an intervention or a waiting control group. Data will be collected before randomisation, after intervention, and after a follow-up of 6 months.

Results

As essential subjects for the curriculum were identified:

* medical background and causes of CRF
* physical activity and moderate exercise
* restructuring daily schedules
* energy conservation
* stress-management and relaxation strategies
* coping with negative emotions
* integrating the new knowledge into every day life.

The program aims at impacting on health-related self-efficacy by the training of problem solving, goal setting, and cognitive techniques as knowledge transfer hasn't proved sufficient to achieve changes in behaviour. According to this we developed a curriculum wherein detailed information for every module concerning objectives, background, didactic methods and materials are provided. Based on the curriculum train-the-trainer seminars are held in order to educate on moderation techniques, group dynamics, and clinical background of CRF. The program will be administered by qualified health professionals in groups of eight patients. It includes six weekly sessions 90 minutes each dealing with the topics listed above.

The results of the pre-test are currently being analysed.

Discussion

Due to the fact that there are no comparable self-management programs for cancer survivors with fatigue the development of the curriculum has been complex. Therefore the critical appraisal by the experts was an important step to validate the program: their contributions have been integrated into the curriculum. The experts appreciated the program as filling in a gap of outpatient cancer care.

ELIGIBILITY:
Inclusion Criteria:

* adult
* malign neoplasms
* ECOG performance status of 0-2
* moderate or severe fatigue
* stable condition after treatment
* German speaking

Exclusion Criteria:

* life expectancy < 1 year
* patients with brain neoplasms
* suicidal tendencies
* severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-01; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Baseline, after the intervention, 6 months later

SECONDARY OUTCOMES:
Quality of Life, Depression and anxiety, physical activity | Baseline, after the intervention, 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Karl Reif, Principal Investigator — IPP

REFERENCES:
- [Derived] Stuhldreher N, Reif K, de Vries U, Gorres S, Petermann F. Development and evaluation of a cancer-related fatigue patient education program: protocol of a randomized controlled trial. BMC Nurs. 2008 Jul 23;7:12. doi: 10.1186/1472-6955-7-12. PMID 18651943